CLINICAL TRIAL: NCT06349551
Title: Clot Formation and Coagulation Factors Consumption Over Time in the Clearing Fluid After Arterial Catheter Blood Sampling in Critically Ill Adult Patients. Prospective Observational Study.
Brief Title: Clot Formation and Coagulation Factors Consumption in the Clearing Fluid After Arterial Catheter Blood Sampling.
Acronym: SECU-BIO2
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC23_0586
Record Dates: First submitted 2024-03-20; First posted 2024-04-05 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Intensive Care Units; Arterial Lines

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Patients of intensive care unit — Patients of intensive care unit having an arterial catheter undergoing arterial blood sampling

SUMMARY:
After blood sampling from an arterial catheter, the reinjection of the clearing fluid (a mixture of saline solution and blood) is proposed to limit blood loss. However, the status of coagulation in this clearing liquid remains poorly documented.

DETAILED DESCRIPTION:
In the intensive care unit, blood sampling is mainly performed through an arterial catheter (radial or femoral artery). In addition to continuous arterial pressure monitoring, this provides an easy access to arterial blood without the need for venipuncture.

It is standard practice to first clear the arterial sampling line before drawing blood for biological tests, to prevent the blood sample from being diluted by the arterial catheter's perfusion solution. This clearing fluid (i.e., a mixture of saline solution and blood) is usually discarded. It has been reported that the clearing fluid volume alone represents 24 to 30% of the total blood volume required for blood sampling.

Devices for reinjecting this clearing fluid are already on the market. The advantages of these devices include blood saving, reduced risk of blood exposure, reduced biological waste and lower infection rates associated with catheter handling. The main drawback of these devices is their cost and the need for frequent replacement. Moreover, their impact on the decrease of blood transfusion remains unclear.

Furthermore, there are too few published data on the potential coagulation of clearing fluid reinjected into the patient nor the maximum time it can be safely reinjected.

The aim of this study is to assess the activation of coagulation over time in the clearing fluid during arterial catheter blood sampling

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years old
* Admitted to the ICU
* With a radial or femoral arterial catheter
* Requiring blood sampling

Exclusion Criteria:

* Presence of a non-standard extension line: any tubing other than an arterial line intended for this purpose.
* Constitutional or acquired hemorrhagic disease,
* Major biological thrombophilia (anti-phospholipid syndrome, homozygous mutation of factor II or V, protein C, S or antithrombin deficiency),
* Thromboembolic event in progress or < 6 months,
* Bacteremia within the last 48 hours,
* Previous study participation,
* Pregnant or breast-feeding patient
* Moribund patient or patient with decision of withholding or withdrawing life-sustaining treatment
* Patient with no health insurance
* Patient under guardianship

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patient with arterial catheter (radial or femoral).
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2024-04-16 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2025-05-21 (Actual)

PRIMARY OUTCOMES:
Composite score of the coagulation activation over time in the clearing fluid during blood sampling from an arterial catheter | 5 minutes (T5)
  Activation of coagulation in the clearing fluid will be assessed by a composite criterion defined by:
  * the presence of a macroscopic clot (binary YES or NO criterion) or
  * fibrinogen consumption (binary YES or NO criterion). Fibrinogen consumption will be classified as YES when its decrease, compared with the reference value measured at T0, is greater than the known technical variability of the assay method

SECONDARY OUTCOMES:
Concentration of prothrombin over time in the clearing fluid during blood sampling from an arterial catheter | 5 minutes (T5)
  Prothrombin time will be assayed at T0, T3 and T5
Concentration of factor II over time in the clearing fluid during blood sampling from an arterial catheter | 5 minutes (T5)
  Factor II will be assayed at T0, T3 and T5
Concentration of factor V over time in the clearing fluid during blood sampling from an arterial catheter | 5 minutes (T5)
  Factor V will be assayed at T0, T3 and T5
Concentration of fibrin monomer over time in the clearing fluid during blood sampling from an arterial catheter | 5 minutes (T5)
  Fibrin monomers will be assayed at T0, T3 and T5

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Nantes university hospital, Nantes, Loire-atlantique
  - Hospital center, Saint-Nazaire